CLINICAL TRIAL: NCT07224698
Title: Phase 2 Multicenter Randomized Placebo-controlled, Double-blind, Parallel Study to Assess the Safety and Efficacy of Inhaled Cannabis in Veterans for Treatment of Posttraumatic Stress Disorder (PTSD)
Brief Title: Inhaled Cannabis for Treatment of PTSD
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Multidisciplinary Association for Psychedelic Studies (Other)
Collaborators: Changemark Research + Evaluation Ltd. (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: MJP2.
Record Dates: First submitted 2025-11-03; First posted 2025-11-05 (Actual); Last update posted 2025-12-10 (Actual); Status verified 2025-12

CONDITIONS: Post Traumatic Stress Disorder PTSD
Keywords: PTSD; Veteran; cannabis; inhaled cannabis; THC; posttraumatic stress disorder; Veteran Affairs
MeSH Terms: conditions — Combat Disorders; Stress Disorders, Post-Traumatic; Marijuana Abuse

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- Active Treatment (Experimental)
  Interventions: Drug: High THC Cannabis
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebo cannabis

INTERVENTIONS:
Drug: High THC Cannabis — dried flower of the Cannabis sativa or indica plant with high (18-22%) THC content
  Arms: Active Treatment
Drug: Placebo cannabis — Placebo contains <1% THC
  Arms: Placebo

SUMMARY:
The rationale for the use of inhalational cannabis to potentially treat PTSD symptoms is based on the many reports of cannabis attenuating PTSD symptom expression among individuals with PTSD, including veterans. Study MJP2 is intended to build off MJP-1 through use of a larger sample size, a parallel study design, and subjective bias mitigation methods to re-examine the use of inhaled high THC-containing cannabis versus placebo for management of PTSD symptoms in a U.S. Veteran sample. Together these studies are intended to provide valuable insights on the already widespread use of cannabis in individuals with PTSD, for which there is currently a lack of controlled evidence available reflective of this real-world use.

ELIGIBILITY:
Inclusion Criteria:

1. Be at least 18 years old.
2. Be a veteran with PTSD lasting 6 months in duration.
3. Meet DSM-5 criteria for PTSD with symptoms (as assessed by the MINI).
4. Have PTSD of at least moderate severity (PCL-5 score of 33 or more) at the time of screening.
5. For participants assigned female sex at birth:

   a) A participant is eligible to participate if not pregnant, and one of the following conditions applies: i) Is not able to become pregnant as defined in protocol (Appendix 2) OR ii) Is a person able to be pregnant (PABP) and using a contraceptive method that is highly effective, with a failure rate of <1%, as described in the protocol (Appendix 2) during the study intervention period and for at least 14 days after the Study Termination visit. The investigator should evaluate the potential for contraceptive method failure (e.g., noncompliance, recently initiated) in relationship to the first dose of study intervention.

   b) A PABP must have a negative highly sensitive pregnancy test (urine or serum as required by local regulations) at Screening, Introductory Session 1, Resupply, and EoT visits c) The investigator is responsible for review of medical history, menstrual history, and recent sexual activity to decrease the risk for inclusion of a participant with an early undetected pregnancy.
6. Be stable on any pre-study medications and/or psychotherapy prior to study entry, agree to inform physician(s)/clinician(s) providing current care about participation in the study, and agree to report any changes in medication or psychotherapy treatment regimen during the study-to-study staff.
7. Have previously inhaled cannabis (e.g. smoked or vaporized cannabis).
8. Be willing to commit to medication dosing and delivery method, to complete evaluation instruments, and attend all study visits.
9. Agree to use only cannabis provided by site staff and agree to required follow up periods for the duration of the study.
10. Agree to keep all cannabis provided by site staff securely stored in the provided lock box and not to share/distribute cannabis to any other individual.
11. Be proficient in reading and writing in English and able to effectively communicate with site staff.
12. Agree not to participate in any other interventional clinical trials during the study.
13. Must agree to inform the investigators within 48 hours of any medical conditions and procedures.
14. Must provide a contact (relative, spouse, close friend or other support person) who is willing and able to be reached by the investigators in the event of a participant becoming suicidal or unreachable.
15. Must be able and willing to record information digitally on a personal device (phone or computer) with internet access.

Exclusion Criteria:

1. Are pregnant, nursing, or are a person able to become pregnant who are not practicing an effective means of birth control.
2. Have current major depressive disorder with primary psychotic features assessed via the Mini-International Neuropsychiatric Interview (MINI).
3. Have current or past DSM-5 diagnosis of eating disorder with active purging, personality disorders, primary psychotic disorder, or bipolar affective disorder type 1 (as assessed with the MINI and the SCID-5-PD).
4. Have current or past DSM-5 diagnosis of dissociative identity disorder, positive family history (first degree relative) of psychotic disorder or bipolar affective disorder type 1 (as assessed by medical history review).
5. Are at high risk of suicide attempt: any participant presenting current serious suicide risk, as determined through psychiatric interview, responses to Columbia Suicide Severity Rating Scale (C-SSRS), and clinical judgment of the investigator will be excluded; however, history of suicide attempts is not an exclusion. Any participant who is likely to require hospitalization related to suicidal ideation and behavior, in the judgment of the investigator, will not be enrolled. Any participant presenting the following on the Baseline/Screening C-SSRS will be excluded:

   1. Suicidal ideation score of 4 or greater within the last month of the assessment at a frequency of once a week or more.
   2. Suicidal ideation score of 5 within the last 6 months of the assessment.
   3. Any suicidal behavior, including suicide attempts or preparatory acts, within the last 6 months. Participants with non-suicidal self- injurious behavior may be included if approved by the Medical Monitor.
6. Would present serious risk to others as established by clinical interview and contact with treating psychiatrist.
7. Have a current moderate (meets 5 of 11 diagnostic criteria per DSM-5) or severe (meets at least 6 of 11 diagnostic criteria per DSM-5) alcohol or cannabis use disorder within the 12 months prior to enrollment. Participants with a substance use disorder other than alcohol or cannabis are excluded.
8. Have a positive urine drug screen for opiates, methamphetamine, cocaine, THC, and amphetamines (unless prescribed). Participants with a positive THC urine analysis tests are excluded from the study but will be allowed to rescreen (maximum twice) after a 1-month cessation of cannabis use.
9. Have a history of arrhythmia, other than occasional premature atrial contractions (PACs) and PVCs in the absence of ischemic heart disease, within 12 months of screening.

   * Participants with a history of atrial fibrillation, atrial tachycardia, atrial flutter or paroxysmal supraventricular tachycardia or any other arrhythmia associated with a bypass tract may be enrolled only if they have been successfully treated with ablation and have not had recurrent arrhythmia for at least one year off all antiarrhythmic drugs, or are under adequate and stable pharmacologic treatment for atrial fibrillation for at least a year, as confirmed by a cardiologist.
10. Have a current or history of chronic obstructive pulmonary disease or asthma.
11. Have a current diagnosis or evidence of significant or uncontrolled hematological, endocrine, cerebrovascular, cardiovascular, coronary, pulmonary, gastrointestinal, renal, hepatic, immunocompromising, or neurological disease according to CI's discretion.
12. Have any current problem, which in the opinion of the CI or Medical Monitor, might interfere with participation.
13. Have any known allergies to cannabis or contraindication for inhalation of cannabis.
14. Are not able to give adequate informed consent.
15. Are not able to attend required face-to-face visits or those who plan to move out of the area within the treatment period.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 320 (Estimated)
Dates: Start 2026-02-01 (Estimated); Primary Completion 2027-06-30 (Estimated); Study Completion 2027-11-30 (Estimated)

PRIMARY OUTCOMES:
Efficacy: Compare changes in PTSD symptom severity in the high THC vs placebo cannabis group as measured by Clinician Administered PTSD Scale for DSM-5, Revised (CAPS-5-R). | Intro 1 (Day 1), End of Treatment (Day 35)
  The CAPS-5 is a 30-item semi-structured interview assessing PTSD in the past month through diagnostic and symptom severity scores anchored to a DSM-5 defined traumatic event. The CAPS-5 produces a Total Severity Score based on severity of PTSD domains described in the DSM-5, as well as a categorical rating indicating whether a participant meets PTSD diagnostic criteria. CAPS-5 Total Symptom Severity scores range from 0 to 80 with higher values indicating greater symptom severity. CAPS-5 assigns PTSD diagnosis as being present or absent.

SECONDARY OUTCOMES:
Compare changes in clinician-rated functional impairment in the high THC vs placebo cannabis group as measured by the Sheehan Disability Scale (SDS). | Intro 1 (Day 1), End of Treatment (Day 35)
  The Sheehan Disability Scale (SDS) is a clinician-rated assessment of functional impairment that was adapted for the purposes of this study to limit missing item-level data as per the FDA requirements and included use of the three-item mean as the total score and imputation of work-related impairment. The SDS is a 3-item scale measuring the severity of disability in the domains of work, family life/home responsibilities and social/leisure activities, with each item scored on a ten-point Likert scale from 0 ('not at all impaired') to 10 ('very severely impaired'). The SDS total score was the mean of the 3 item responses. The SDS total score ranged from 0 to 10, with higher scores indicating greater functional impairment.

CONTACTS AND LOCATIONS:
Locations (1):
- Scottsdale Research Institute, Cave Creek, Arizona, United States

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- See also: Related Info — https://maps.org/marijuana/mjp2/